CLINICAL TRIAL: NCT03897478
Title: Biomarkers of Acute Stroke in Clinic
Acronym: BASIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ischemia Care LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: NCT02014896-2
Record Dates: First submitted 2019-03-25; First posted 2019-04-01 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Ischemic Stroke; Ischemia; Atrial Fibrillation; Transient Ischemic Attack; Transient Cerebrovascular Events; Thrombotic Stroke; Stroke; Stroke, Acute; Stroke, Ischemic; Stroke, Complication; Stroke of Basilar Artery; Atherosclerosis; Atheroma; Cardioembolic Stroke; Cardiomyopathies; Cardiovascular Stroke; Thromboembolism
Keywords: Ischemic stroke; Atrial fibrillation; Transient neurological event; Cryptogenic stroke; Gene expression; RNA; Anticoagulant; NOAC; Implantable cardiac monitor; Point of care; tPA; Thrombectomy; Cardiac monitoring
MeSH Terms: conditions — Ischemic Stroke; Ischemia; Atrial Fibrillation; Ischemic Attack, Transient; Thrombotic Stroke; Stroke; Atherosclerosis; Plaque, Atherosclerotic; Embolic Stroke; Cardiomyopathies; Myocardial Infarction; Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biospecimen will be whole blood samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ischemic Stroke: Ischemic stroke subjects presenting within 30 hours from symptom onset will have al PAX Gene Blood RNA tubes drawn upon arrival to the Emergency Department (if available) or hospital.
  Biomarker blood draw
  Interventions: Diagnostic Test: ISCDX blood test
- Control: Control group subjects will have PAX Gene Blood RNA tubes drawn. Control group matched with ischemic stroke subjects for age, race, gender, smoking history with at least one of the following vascular risk factors: diabetes, hypertension, atrial fibrillation, hyperlipidemia.
  Biomarker blood draw

INTERVENTIONS:
Diagnostic Test: ISCDX blood test — The ISCDX test is based on gene expression changes that occur as a result of the ischemic stroke. When the stroke occurs, the immune system in the body reacts and causes changes in gene expression in several types of cells, including white blood cells, related to activation of innate and adaptive immune systems.
  The ISCDX test distinguishes between cardioembolic and large artery atherosclerotic origin of stroke using a gene signature. The pattern or signature of up or down regulation for all genes for a patient determines whether the patient's pattern of gene expression is more like the pattern seen in other cardioembolic patients or more like the pattern seen in patients with large artery atherosclerotic cause of stroke.
  Groups: Ischemic Stroke

SUMMARY:
The proposed study will investigate the clinical use of the ISCDX test that may differentiate between diverse stroke etiologies as listed below:

Aim 1: Differentiate between cardioembolic and large artery atherosclerotic ischemic strokes, when hemorrhagic stroke is ruled out, as defined by TOAST classification of subtypes of acute ischemic stroke.

Aim 2: In cases of ischemic strokes of unknown or "cryptogenic" etiology, determine the ability of biomarker blood tests to predict etiology between cardioembolic and large artery atherosclerotic.

DETAILED DESCRIPTION:
Acute ischemic stroke (AIS) is a leading cause of adult mortality and morbidity in the United States, affecting over 800,000 individuals, annually, leaving many with permanent disability. Emergent evaluation, prompt acute treatment, and identification of stroke etiology for secondary prevention are key to decreasing the morbidity and mortality associated with cerebrovascular disease. Key to treatment and prevention is the identification of stroke etiology - large vessel atherosclerosis, cardioembolic phenomenon, or in-situ small vessel cerebrovascular disease - since primary and secondary prevention measures differ based on stroke subtype. The diagnosis of ischemic stroke includes a combination of patient history, clinical assessment, and brain imaging. However, identifying the cause of cerebrovascular ischemia is challenging and routinely assigned of cryptogenic origin.

Therefore, the need is great, to understand the pathogenesis of AIS events in order to develop more effective preventative measures. Recent studies have identified the differential expression of genes in whole blood which may differentiate the major ischemic stroke types. Such differences may help identify AIS events that are more likely to respond to therapy specifically tailored to the major stroke type. Furthermore, by establishing a more robust standard for secondary prevention, future stroke events may be avoided.

BASIC is a multisite prospective study with a estimated enrollment of up to 500 consecutive adult subjects including no more than 50 age, gender and co-morbidity matched controls ("Controls"). Stroke subjects will be recruited from patients who present to the Emergency Department (ED) or hospital with suspected AIS. Research personnel will identify potential patients by responding to "Brain Attack" pages from the ED to the Stroke Team for patients who meet current Brain Attack criteria. Following evaluation by the ED and neurology physicians, the clinical coordinator will verify the patient had a suspected AIS and meets eligibility criteria. The patient or their legal surrogate will be approached for study participation. Written informed consent will be obtained for all subjects enrolled.

Control subjects will be those who present to the Emergency Department for non-stroke reasons but have one or more risk factors for stroke. These subjects will not have a recruitment window. They can be consented as they present to the hospital. Tubes will be marked as controls. In past studies, these have been collected during slow times in the Emergency Department. Once the study has reached 50 controls, the sponsor will stop enrolling for this group. This has been done in the past by sending the sites a communication that the control group quota has been reached.

The recruitment window will be determined by time of symptom onset, time of presentation at ED or hospital, and ability to consent. This will include patients that present within 30 hours of symptom onset or last known normal time and clinical evidence suggesting Acute Ischemic Stroke.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 and < 80 years of age.
* Signs and symptoms suggestive of AIS due to cardioembolic, large vessel, or unknown etiology according to TOAST criteria.
* Arrival to the ED within 30 hours of symptom onset or last known normal time and clinical evidence suggesting Acute Ischemic Stroke.
* Head CT or MRI ruling out other pathology such as vascular malformation, hemorrhage, tumor or abscess which would likely be responsible for presenting neurologic symptoms
* Informed consent obtained

Exclusion Criteria:

* Any central nervous system infection, i.e. meningitis or encephalitis in the past 30 days
* Any form of head trauma, stroke or intracranial hemorrhage in the past 30 days
* Any history of primary or metastatic brain cancer
* Active cancer defined as a diagnosis of cancer, within 6 months before enrollment, any treatment for cancer within the previous 6 months, or recurrent or metastatic cancer.
* Autoimmune diseases: such as lupus, rheumatoid arthritis, Crohn's disease, ulcerative colitis
* Active chronic infectious diseases (eg. HIV/AIDS, hepatitis C)
* Any underlying medical condition which in the opinion of the investigator would prohibit the patient from providing informed consent
* Major surgery within three months prior to the index event
* Signs and symptoms suggestive of (i) AIS due to small vessel occlusion (lacune) and other known etiology according to TOAST criteria, as well as (ii) stroke mimics, transient ischemic attacks, or transient neurological events.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Source of Subject Population:
  Ischemic stroke population will be adult patients who present to the Emergency Department or hospital with an acute ischemic strokeor meet the definition of a control subject who meet the inclusion/exclusion criteria.
  Controls subjects will be non-neurologic patients who are matched with the stroke patients for age, race, gender and smoking plus one or more of the following co-morbidities or vascular risk factors:
  1. Diabetes
  2. Hypertension
  3. Atrial fibrillation
  4. Hyperlipidemia
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of the rates of patients presenting with acute ischemic stroke identified with ISCDX testing with TOAST criteria | up to 1 year
  The ISCDX test results will be compared to acute ischemic stroke assessment as defined by the TOAST criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio Health Riveside Methodist Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jauch EC, Barreto AD, Broderick JP, Char DM, Cucchiara BL, Devlin TG, Haddock AJ, Hicks WJ, Hiestand BC, Jickling GC, June J, Liebeskind DS, Lowenkopf TJ, Miller JB, O'Neill J, Schoonover TL, Sharp FR, Peacock WF. Biomarkers of Acute Stroke Etiology (BASE) Study Methodology. Transl Stroke Res. 2017 May 5;8(5):424-8. doi: 10.1007/s12975-017-0537-3. Online ahead of print. PMID 28477280